CLINICAL TRIAL: NCT02381262
Title: Fitbit / Healthy Weight Management Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Collaborators: Louise von Hess Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-201
Record Dates: First submitted 2015-02-24; First posted 2015-03-06 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Fitbit
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): At the 2 week post-surgical visit, subjects will receive and be trained in the use of the Fitbit and data interface and meet with the exercise physiologist or research coordinator to initiate MyLGHealth, lifestyle/activity data collection.
  Subsequent data collection time-points correspond with follow-up post-surgical appointments either at each visit or the 2 week, 1 month, 4 month, 8 month or 12 month visit.
  Interventions: Behavioral: Fitbit
- Control (No Intervention): At the 2 week post-surgical visit, all subjects will then meet with the exercise physiologist or research coordinator to initiate MyLGHealth, lifestyle/activity data collection.
  Subsequent data collection time-points correspond with follow-up post-surgical appointments either at each visit or the 2 week, 1 month, 4 month, 8 month or 12 month visit.
  The control group will receive a current version of the Fitbit device at the end of their completion of the 12 month visit.
- Historical Control (No Intervention): The investigators will extract historical control data from the electronic health record using electronic queries and manual data extraction. Historical controls will have surgery and 12-month follow-up completed prior to the start of the RCT.

INTERVENTIONS:
Behavioral: Fitbit — The Fitbit is a wrist based wearable technology device designed to monitor physical activity by tracking steps, distance and calories burned as well as sleep patterns and heart rate. It has wireless capabilities to sync with smart devices and summarize data for the user or export for synchronize with electronic health records.
  Arms: Intervention

SUMMARY:
Study Aims Specifically with our Healthy Weight Management patients that are pursuing sleeve gastrectomy surgery, the investigators would like to determine if the Fitbit is associated with health outcomes in this population.

Primary Outcome

• Percentage of excess weight loss - Does the use of a Fitbit positively affect the percentage of excess body weight loss in vertical sleeve gastrectomy patients?

Secondary Outcomes

* Lifestyle changes and Exercise patterns - Does the use of a Fitbit foster positive lifestyle and exercise pattern changes in post-operative VSG patients?
* Resolution of comorbidity - Does the use of a Fitbit positively affect patient health via reduction of co-morbid conditions associated with morbid obesity following VSG surgery?

DETAILED DESCRIPTION:
Study Aims Specifically with our Healthy Weight Management patients that are pursuing sleeve gastrectomy surgery, the investigators would like to determine if the Fitbit is associated with health outcomes in this population.

Primary Outcome

• Percentage of excess weight loss - Does the use of a Fitbit positively affect the percentage of excess body weight loss in vertical sleeve gastrectomy patients?

Secondary Outcomes

* Lifestyle changes and Exercise patterns - Does the use of a Fitbit foster positive lifestyle and exercise pattern changes in post-operative VSG patients?
* Resolution of comorbidity - Does the use of a Fitbit positively affect patient health via reduction of co-morbid conditions associated with morbid obesity following VSG surgery?

Research Methodology This study will be focused on a bariatric post-surgical population and is designed as a randomized controlled trial (RCT) with three arms; a RCT with a control and intervention group and a historical control group. For the RCT, subjects, after providing informed consent, will be randomized into either the control arm or the intervention arm. In the control arm, subjects will be provided normal/standard of care for post-surgical bariatric patients. This includes physician visits, dietary and exercise consults, education and other therapy as appropriate for their care. In the intervention arm, subjects will be provided with a Fitbit bracelet and software to monitor their physical activity in addition to the normal/standard of care provided in the control group. Both groups will receive the recommended aerobic and strength training exercise guidelines. Furthermore, each group will have identical exercise education regarding appropriate intensity using either rate of perceived exertion or target heart rate range. At the end of the 12-month tracking period of the study, the control group will be provided with a Fitbit bracelet so that they can begin tracking their activity levels during the 2nd post-operative year. A third group, the historical controls, at the end of the study will be extracted from the electronic medical records from patients who have meet the same inclusion/exclusion criteria and were surgical patients with completed follow-up prior to the start of the RCT portion of the trial.

RCT subjects randomized to the intervention group will be provided with step by step instructions on how to set-up the Fitbit app on their smartphone and or view the data on the Fitbit secure portal. Additionally, subjects will be shown how to track their weekly structured aerobic and strength training exercise within the app. Users will also be shown how to access Fitbit data on the MyLGHealth portal. Data from the Fitbit will also be accessible to the provider on EPIC flow sheets. Providers will be able to incorporate this data into discussions with patient at visits. RCT subjects randomized to the control group will receive the same training and a Fitbit device after they complete their 12 month visit.

Just prior to the start of the RCT, we will be conducting a pilot study to test the implementation of the Fitbit in this patient population. The pilot phase will initially target 5 patients to enroll as a test of the set-up of the Fitbit monitoring, data transfer, activity logs and other data collection procedures. Subjects in this pilot phase will only participate for a period of 1 month and all individuals will receive a Fitbit device. The investigators will employ all inclusion/exclusion criteria, recruitment procedures and complete all data collection procedures (baseline and follow-up) as planned for the randomized trial. If additional adjustments need to be made relative to the Fitbit set-up or training/reference materials for patients, another 5 pilot patients may be recruited. Data collection and study procedures on all pilot subjects will be completed before the randomized trial begins. This pilot study will be submitted to the IRB for review and approval as a separate study prior to the RCT portion of the study.

For the RCT portion of the study, subjects will be recruited, enrolled and randomized into the study and then baseline data will be collected and entered into the study database. These data elements include subject demographics (age, gender, weight entering program, preoperative weight, comorbidities, lifestyle and physical activity patterns, etc.). Subjects will be followed for one year or until lost to follow-up with data collected at each physician office visit. At each office visit, the investigators will extract from Epic the date of the visit, subject weight and comorbidities. Lifestyle and physical activity patterns will only be assessed at the 2 week, 1 month, 4 month, 8 month and 12 month visits. The historical control group will be extracted at the end of the study when RCT subjects are nearing the completion of their 12 month follow-up.

The historical controls will consist of a group of patients that will have already received surgery and completed 12 month follow-up prior to the start of the pilot and RCT portions of the project. There will be no interaction with them as a part of the study. The investigators are planning to identify them and collect data at the end of the RCT portion of the project.

ELIGIBILITY:
Inclusion Criteria:

* Naive bariatric surgery procedure patients - approved for surgery
* Laparoscopic VSG patients
* Completion of all pre-surgical requirements
* Age ≥ 18
* Subject must have a My LG Health account activated
* Subject must have a PC and/or Bluetooth enabled device at home

Exclusion Criteria:

* Band procedures
* Revisions
* All other bariatric procedures
* Non-English speaking patient (justification - My LG Health information and support is only available in English)
* Already own and use a Fitbit type device
* Cognitive impairments or lack of support that would limit the abilities to comply with study procedures or use of a diary/Fitbit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of excess weight loss | 1 year
  Does the use of a Fitbit positively affect the percentage of excess body weight loss in VSG patients?
  Subjects enrolled in the study will have ideal body weight (IBW) calculated upon entry into the bariatric program and entered into the electronic health record. IBW calculations are based on the Met Life IBW charts. EWL at the end of one year will be calculated as follows:
  EWL% = (ABW - CW)/EBW *100 EWL%: Percentage of excess weight loss CW: Current weight (to be collected at regular intervals during the study, but for purposes of this objective, the measure collected at the 1 year visit) ABW: Actual body weight at baseline - date approved for surgery and entering pre-surgical period EBW: Excess body weight = ABW - IBW IBW: Ideal body weight based on Met Life IBW charts

SECONDARY OUTCOMES:
Changes and physical activity patterns | 1 year
  Does the use of a Fitbit foster positive physical activity pattern changes in post-operative VSG patients?
  Subjects will complete the International Physical Activity Questionnaire (IPAQ-LF) long form which consists of questions to assess physical activity over the past 7 days. The IPAQ will be administered at regular office visits to both the control and intervention groups at 2 weeks, 1 month, 4 months, 8 months, 1 year follow-up visits.
Resolution of comorbidity | 1 year
  Does the use of a Fitbit positively affect patient health via reduction of co-morbid conditions associated with morbid obesity following VSG surgery?
  Subjects in all three groups will have standard comorbidity assessments for the following diseases:
  * Diabetes, based on number of diabetes medications and HA1C of 6.5
  * Hypertension, based on number of antihypertensives
  * Hyperlipidemia, based on number of lipid lowering medications and total cholesterol or triglyceride level of 200
  * Obstructive sleep apnea, based on use of CPAP or BiPAP These assessments will occur at baseline and at the 2 weeks, 1 month, 4 months, 8 months, 1 year follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: James Ku, MD, Principal Investigator — Lancaster General Bariatric Surgery and Healthy Weight Management Programs
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anton SD, LeBlanc E, Allen HR, Karabetian C, Sacks F, Bray G, Williamson DA. Use of a computerized tracking system to monitor and provide feedback on dietary goals for calorie-restricted diets: the POUNDS LOST study. J Diabetes Sci Technol. 2012 Sep 1;6(5):1216-25. doi: 10.1177/193229681200600527. PMID 23063049
- [Background] Burke LE, Styn MA, Sereika SM, Conroy MB, Ye L, Glanz K, Sevick MA, Ewing LJ. Using mHealth technology to enhance self-monitoring for weight loss: a randomized trial. Am J Prev Med. 2012 Jul;43(1):20-6. doi: 10.1016/j.amepre.2012.03.016. PMID 22704741
- [Background] Carter MC, Burley VJ, Nykjaer C, Cade JE. Adherence to a smartphone application for weight loss compared to website and paper diary: pilot randomized controlled trial. J Med Internet Res. 2013 Apr 15;15(4):e32. doi: 10.2196/jmir.2283. PMID 23587561
- [Background] Chambliss HO, Huber RC, Finley CE, McDoniel SO, Kitzman-Ulrich H, Wilkinson WJ. Computerized self-monitoring and technology-assisted feedback for weight loss with and without an enhanced behavioral component. Patient Educ Couns. 2011 Dec;85(3):375-82. doi: 10.1016/j.pec.2010.12.024. Epub 2011 Feb 3. PMID 21295433
- [Background] Conroy MB, Yang K, Elci OU, Gabriel KP, Styn MA, Wang J, Kriska AM, Sereika SM, Burke LE. Physical activity self-monitoring and weight loss: 6-month results of the SMART trial. Med Sci Sports Exerc. 2011 Aug;43(8):1568-74. doi: 10.1249/MSS.0b013e31820b9395. PMID 21200337
- [Background] Cook DJ, Thompson JE, Prinsen SK, Dearani JA, Deschamps C. Functional recovery in the elderly after major surgery: assessment of mobility recovery using wireless technology. Ann Thorac Surg. 2013 Sep;96(3):1057-61. doi: 10.1016/j.athoracsur.2013.05.092. PMID 23992697
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Manzoni GM, Pagnini F, Corti S, Molinari E, Castelnuovo G. Internet-based behavioral interventions for obesity: an updated systematic review. Clin Pract Epidemiol Ment Health. 2011 Mar 4;7:19-28. doi: 10.2174/1745017901107010019. PMID 21552423
- [Background] Morgan PJ, Callister R, Collins CE, Plotnikoff RC, Young MD, Berry N, McElduff P, Burrows T, Aguiar E, Saunders KL. The SHED-IT community trial: a randomized controlled trial of internet- and paper-based weight loss programs tailored for overweight and obese men. Ann Behav Med. 2013 Apr;45(2):139-52. doi: 10.1007/s12160-012-9424-z. PMID 23129021
- [Background] Mundi MS, Lorentz PA, Swain J, Grothe K, Collazo-Clavell M. Moderate physical activity as predictor of weight loss after bariatric surgery. Obes Surg. 2013 Oct;23(10):1645-9. doi: 10.1007/s11695-013-0979-y. PMID 23636999
- [Background] Adam Noah J, Spierer DK, Gu J, Bronner S. Comparison of steps and energy expenditure assessment in adults of Fitbit Tracker and Ultra to the Actical and indirect calorimetry. J Med Eng Technol. 2013 Oct;37(7):456-62. doi: 10.3109/03091902.2013.831135. Epub 2013 Sep 5. PMID 24007317
- [Background] Reames BN, Finks JF, Bacal D, Carlin AM, Dimick JB. Changes in bariatric surgery procedure use in Michigan, 2006-2013. JAMA. 2014 Sep 3;312(9):959-61. doi: 10.1001/jama.2014.7651. No abstract available. PMID 25182106
- [Background] Shada AL, Hallowell PT, Schirmer BD, Smith PW. Aerobic exercise is associated with improved weight loss after laparoscopic adjustable gastric banding. Obes Surg. 2013 May;23(5):608-12. doi: 10.1007/s11695-012-0826-6. PMID 23196991
- [Background] Shuger SL, Barry VW, Sui X, McClain A, Hand GA, Wilcox S, Meriwether RA, Hardin JW, Blair SN. Electronic feedback in a diet- and physical activity-based lifestyle intervention for weight loss: a randomized controlled trial. Int J Behav Nutr Phys Act. 2011 May 18;8:41. doi: 10.1186/1479-5868-8-41. PMID 21592351
- [Background] Sjostrom CD, Lissner L, Wedel H, Sjostrom L. Reduction in incidence of diabetes, hypertension and lipid disturbances after intentional weight loss induced by bariatric surgery: the SOS Intervention Study. Obes Res. 1999 Sep;7(5):477-84. doi: 10.1002/j.1550-8528.1999.tb00436.x. PMID 10509605
- [Background] Smith BR, Schauer P, Nguyen NT. Surgical approaches to the treatment of obesity: bariatric surgery. Endocrinol Metab Clin North Am. 2008 Dec;37(4):943-64. doi: 10.1016/j.ecl.2008.08.001. PMID 19026941
- [Background] Thompson WG, Kuhle CL, Koepp GA, McCrady-Spitzer SK, Levine JA. "Go4Life" exercise counseling, accelerometer feedback, and activity levels in older people. Arch Gerontol Geriatr. 2014 May-Jun;58(3):314-9. doi: 10.1016/j.archger.2014.01.004. Epub 2014 Jan 15. PMID 24485546
- [Background] Turk MW, Elci OU, Wang J, Sereika SM, Ewing LJ, Acharya SD, Glanz K, Burke LE. Self-monitoring as a mediator of weight loss in the SMART randomized clinical trial. Int J Behav Med. 2013 Dec;20(4):556-61. doi: 10.1007/s12529-012-9259-9. PMID 22936524
- [Background] Unick JL, O'Leary KC, Bond DS, Wing RR. Physical activity enhancement to a behavioral weight loss program for severely obese individuals: A preliminary investigation. ISRN Obes. 2012 Sep 5;2012:465158. doi: 10.5402/2012/465158. PMID 24379985
- [Background] Wang J, Sereika SM, Chasens ER, Ewing LJ, Matthews JT, Burke LE. Effect of adherence to self-monitoring of diet and physical activity on weight loss in a technology-supported behavioral intervention. Patient Prefer Adherence. 2012;6:221-6. doi: 10.2147/PPA.S28889. Epub 2012 Mar 22. PMID 22536058